CLINICAL TRIAL: NCT01002820
Title: A Treatment Protocol for Ganaxolone as add-on Therapy in Adult Patients With Uncontrolled Partial-onset Seizures Deriving Benefit From Protocol 1042-0601
Brief Title: A Treatment Use Protocol for Subjects Continuing on From the Open-label Extension 0601
Acronym: 0602
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1042-0602
Record Dates: First submitted 2009-10-16; First posted 2009-10-27 (Estimated); Results first posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-05

CONDITIONS: Epilepsy, Complex Partial
Keywords: Epileptic Seizures; Seizure Disorder; Seizures; Convulsions; Anticonvulsant; Anticonvulsive; Antiepileptic; Ganaxolone
MeSH Terms: conditions — Epilepsy, Complex Partial; Seizures; Epilepsy | interventions — ganaxolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- participants (Experimental): all subjects participating in 0602 are receiving ganaxolone for seizure control
  Interventions: Drug: ganaxolone

INTERVENTIONS:
Drug: ganaxolone — liquid suspension, 50 mg/mL, up to 500 mg/day TID or 1500 mg/day, up to 1 year
  Other Names: CCD 1042; CAS 383-98323-2; 3 alpha-hydroxy, 3 beta-methyl, 5 alpha-pregnan-20-one

SUMMARY:
This study is designed to provide ganaxolone to those patients deriving significant benefit from current treatment in protocol 1042-0601.

ELIGIBILITY:
Inclusion Criteria:

* subjects who have completed all study visits from previous protocol 1042-0601 and have been deemed eligible by the Investigator as:
* having had no major adverse events thought to be drug related
* deriving benefit from ganaxolone treatment
* be properly informed of the nature and risks of the study and give written informed consent prior to study entry
* must be willing to use a medically acceptable method of birth control and if female of child-bearing potential, have a negative qualitative serum pregnancy test

Exclusion Criteria:

* significant medical or surgical condition at screening or that develops during protocol participation that might compromise hematologic, cardiovascular, pulmonary, renal, gastrointestinal, or hepatic systems, or other conditions that would place the subject under increased risk
* unwilling to use a double-barrier method of birth control or submit to a serum pregnancy test
* history of chronic non-compliance with drug regimens
* females currently breastfeeding
* AST or ALT levels greater than 3 times the upper limit of normal at screen
* Inability to withhold grapefruit or grapefruit products during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Southern California, Dept of Neurology, Los Angeles, California
  - University of Kentucky, Dept of Neurology, Lexington, Kentucky
  - Albany Medical Center, Dept of Neurology, Albany, New York
  - Ohio State University, Columbus, Ohio
  - Riddle Health Care Center II, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Comprehensive Epilepsy Center, Philadelphia, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population was to have completed all scheduled clinical study visits in the previous protocol 1042-0601 and have been deemed eligible by the Investigator including no major adverse events [AEs] thought to be drug related and deriving benefit from ganaxolone treatment.
Period: Overall Study
Arm/Group | Ganaxolone
Started | 11
Completed | 7
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: ITT Population
Arm/Group | Ganaxolone
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Investigators Global Assessment
Description: Investigator's global assessment of the patient's response to ganaxolone treatment was collected during the study to support continued trial participation. The investigator's global assessment of the patient's response to ganaxolone treatment was collected during the study to support continued trial participation. Responses categories were Improved Markedly, Improved Moderately, Improved Slightly and No change from baseline.
Time Frame: Screening through 52 weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone
Number analyzed (Participants) | 11
Participants
  Improved Markedly - Visit 1 - Screening | 6
  Improved Moderately - Visit 1 - Screening | 4
  Improved Slightly - Visit 1 - Screening | 0
  No change from baseline - Visit 1 - Screening | 1
  Improved Markedly - Visit 2 - Week 26: number analyzed (Participants) | 7
  Improved Markedly - Visit 2 - Week 26 | 3
  Improved Moderately - Visit 2 - Week 26: number analyzed (Participants) | 7
  Improved Moderately - Visit 2 - Week 26 | 4
  Improved Slightly - Visit 2 - Week 26: number analyzed (Participants) | 7
  Improved Slightly - Visit 2 - Week 26 | 0
  No change from baseline - Visit 2 - Week 26: number analyzed (Participants) | 7
  No change from baseline - Visit 2 - Week 26 | 0
  Improved Markedly - Visit 3 - Week 52 or Taper Visit: number analyzed (Participants) | 8
  Improved Markedly - Visit 3 - Week 52 or Taper Visit | 2
  Improved Moderately - Visit 3 - Week 52 or Taper Visit: number analyzed (Participants) | 8
  Improved Moderately - Visit 3 - Week 52 or Taper Visit | 4
  Improved Slightly - Visit 3 - Week 52 or Taper Visit: number analyzed (Participants) | 8
  Improved Slightly - Visit 3 - Week 52 or Taper Visit | 1
  No change from baseline - Visit 3 - Week 52 or Taper Visit: number analyzed (Participants) | 8
  No change from baseline - Visit 3 - Week 52 or Taper Visit | 1

ADVERSE EVENTS:
Time Frame: Screening (0601 visit 12/last visit) through Visit 4 (week 56 - last visit)
Arm/Group | Ganaxolone
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=11)
Tension headache (Nervous system disorders) | 1
Transient ischemic attack (Nervous system disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=11)
Diarrhea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Irritability (General disorders) | 2
Fatigue (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Nail Tinea (Infections and infestations) | 1
Tinea Pedis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 2
Complex Partial Seizures (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Intracranial Aneurysm (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tension Headache (Nervous system disorders) | 1
Transient Ischaemic Attack (Nervous system disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1
Aortic Aneurysm (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Efficacy measurements were not collected in this study. The investigator's global impression was recorded to justify continued ganaxolone treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No